CLINICAL TRIAL: NCT04754672
Title: Aerobic Fitness or Muscle Mass Training to Improve Colorectal Cancer Outcome (AMICO). The Effects of Exercise on Chemotherapy Dose Modification and Progression Free Survival in Patients With Metastatic Colorectal Cancer
Brief Title: Aerobic Fitness or Muscle Mass Training to Improve Colorectal Cancer Outcome
Acronym: AMICO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: UMC Utrecht (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Rijnstate Hospital (Other); Jeroen Bosch Ziekenhuis (Other); Flevoziekenhuis (Other); Catharina Ziekenhuis Eindhoven (Other); Meander Medical Center (Other); Ziekenhuis Amstelland (Other); Amphia Hospital (Other); Spaarne Gasthuis (Other); Canisius-Wilhelmina Hospital (Other); Amsterdam UMC, location VUmc (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-6867; NL72482.091.20 (Other: CCMO); 09150171910017 (Other Grant/Funding Number: NWO-VIDI)
Record Dates: First submitted 2020-12-04; First posted 2021-02-15 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer; Chemotherapeutic Toxicity; Survivorship; Lifestyle
Keywords: Exercise; Muscle strength; Cardiorespiratory fitness; Colorectal cancer; Chemotherapy dose modification; Progression free survival; Bayesian adaptive trial
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Masking Description: Treatment allocation is concealed. Baseline assessments prior to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continuous aerobic and resistance exercise (AE+RE) (Experimental): Two 60 min moderate-to-high intensity exercise sessions per week supervised by a physiotherapist.
  Continuous aerobic exercise: 15-20 min continuous aerobic exercise (e.g. walking) of moderate intensity (Borg 13-14 'somewhat hard').
  Resistance exercise (25 min): 6 exercises targeting large muscle groups vertical row, squat, bench press, pull over, abdominal crunch, and lunge. 2 sets of 10 repetitions at 70-80% of 1 RM. To ensure adequate training load over time, tests are repeated every 3/4 weeks aligned with the chemotherapy cycle.
  One additional (third) session from home at moderate intensity for at least 30 min.
  A brochure with exercise guidelines is provided.
  Interventions: Behavioral: Continuous aerobic and resistance exercise intervention
- Continuous aerobic and aerobic interval exercise (AE+AI) (Experimental): Continuous aerobic exercise: 15-20 min continuous aerobic exercise (e.g. walking) of moderate intensity (Borg 13-14 'somewhat hard').
  Aerobic interval (25 min): cycling with high intensity intervals alternated with recovery intervals. Intensity of the interval: between 85% and 95% of estimated maximum heart rate, adjusted to Borg 16-18 'hard - very hard'. In between the intervals, light intensity cycling will be performed for active recovery at 30% of Wmax estimated from Steep ramp test and adjusted to Borg < 12.
  One additional (third) session from home at moderate intensity for at least 30 min.
  A brochure with exercise guidelines is provided.
  Interventions: Behavioral: Continuous aerobic and aerobic interval exercise intervention
- Usual care control group (No Intervention): Patients in the usual care group receive care as usual. In addition, a brochure with exercise guidelines for cancer survivors is provided

INTERVENTIONS:
Behavioral: Continuous aerobic and resistance exercise intervention — Continuous aerobic and resistance exercises intervention
  Other Names: AE+RE
  Arms: Continuous aerobic and resistance exercise (AE+RE)
Behavioral: Continuous aerobic and aerobic interval exercise intervention — Continuous aerobic and aerobic interval exercise intervention
  Other Names: AE+AI
  Arms: Continuous aerobic and aerobic interval exercise (AE+AI)

SUMMARY:
Evidence from randomized controlled trials shows that exercise during cancer treatment benefits physical fitness, fatigue and quality of life. Since the effect of exercise on clinical outcome is currently unknown, exercise is not included as integral part of standard cancer care. Moreover, evidence regarding the optimal exercise prescription in terms of type and dose is lacking.

To maintain quality of life in patients receiving palliative treatment with chemotherapy, toxicity-induced modifications in the prescribed chemotherapy dose are common. Such modifications - occurring in 40% of patients with metastatic colorectal cancer - may reduce benefit of treatment. The investigators hypothesize that exercise prevents chemotherapy dose modifications by reducing toxicity and enhancing psychological strength. Additionally, based on studies in rodents and preliminary data in patients with cancer, the researchers hypothesize that exercise has beneficial effects on the functionality of the natural killer cells, which play an important role in the innate immune defense against cancer. Both, fewer dose modifications and improved immune function may improve progression-free survival.

This study is a three-armed trial comparing resistance exercise, aerobic interval exercise and usual care in patients with metastatic colorectal cancer to select the optimal exercise prescription for preventing chemotherapy dose modifications. The trial will use a Bayesian adaptive multi-arm multi-stage design with several interim analyses after which an ineffective study arm can be dropped early. This novel design makes the trial more efficient and reduces patients' exposure to suboptimal study arms.

Evidence regarding the exercise effects on i) clinical outcome, ii) the optimal exercise prescription, and iii) the underlying mechanisms, elucidates the potential of exercise to boost benefit from chemotherapy treatment. This evidence provides leads to improve progression-free survival and quality of life of patients suffering from one of the leading causes of cancer death worldwide.

DETAILED DESCRIPTION:
First-line treatment of metastatic colorectal cancer (mCRC) generally includes the chemotherapies fluoropyrimidines in combination with oxaliplatin and/or irinotecan, known as doublet or triplet chemotherapy. A previous study showed that over 40% of patients with metastatic colorectal cancer required dose modifications (including dose reductions, treatment delays or discontinuation) within the first three months of palliative treatment, and around 30% was admitted to hospital due to chemotherapy-related toxicity. Toxicity-induced dose modifications and hospitalization may reduce benefit of treatment. In patients with metastatic colorectal cancer, reductions in muscle mass and lower physical activity levels (<9 metabolic equivalent of task hours/week) were found to be associated with more dose-limiting toxicity and shorter (progression-free) survival. However, the causality and underlying mechanisms linking physical activity and exercise to cancer outcome have not been elucidated. The immune system (by increased infiltration of activated natural killer cells into the tumour) might play a role as was shown in studies with rodents. In addition, studies among patients showed that exercise may counteract a variety of treatment toxicities (e.g. neutropenia, neuropathy, gastrointestinal side effects, fatigue), but optimal exercise type and dose are unknown.

In addition to the above-mentioned biophysiological effects by which exercise may prevent dose modifications, several studies demonstrated the positive effects of exercise during cancer treatment on quality of life. A recent study on patients' perceptions indicated that exercise helped patients to better cope with cancer treatments, as it gave them psychological strength (i.e. empowerment and resilience) next to physical strength. The investigators hypothesize that exercise reduces treatment-related toxicity and thereby reduces chemotherapy dose modifications and improves progression free survival.

randomised controlled trials are the gold standard for ascertaining treatment efficacy. Studying differences in effects on chemotherapy dose modifications between different exercise programs requires a multi-arm randomised controlled trial. Due to complex logistics and high costs, the conduct of a traditional adequately powered multi-arm exercise trial is difficult with available patients and resources. Therefore, a Bayesian adaptive flexible multi-arm multi-stage design will be used which allows for a number of interim analyses after which a treatment arm can be dropped early if it falls outside the pre-defined futility/efficacy boundaries. This reduces patients' exposure to suboptimal interventions and increases trial efficiency.

This study aims to examine whether:

1. Exercise prevents chemotherapy dose modifications via reduced toxicity and enhanced psychological strength, and which exercise program yields largest benefits.
2. Exercise improves immune function (e.g. functionality of natural killer cells).
3. Benefits of exercise on dose modifications and immune function improves progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* mCRC with indication for palliative chemotherapy
* scheduled for treatment with first-line doublet or triplet chemotherapy, according to the national guideline
* able and willing to give written informed consent.

Exclusion Criteria:

* life expectancy <6 months
* unable to perform basic activities of daily living such as walking or biking
* presence of cognitive disorders or severe emotional instability (e.g., Schizophrenia, Alzheimer, alcohol addiction);
* presence of other disabling co-morbidities that might hamper physical exercise (e.g. heart failure (NYHA classes 3 and 4), chronic obstructive pulmonary disease (COPD, gold 3 and 4), orthopaedic conditions and neurological disorders (e.g., hernia, paresis, amputation, active rheumatoid arthritis);
* insufficient mastery of the Dutch language;
* presence of serious cardiovascular or cardiopulmonary conditions (e.g. unstable angina, arrhythmia or valve disease) such that exercise safety is at risk, as judged by the treating physician.
* Already participating in structured vigorous aerobic and/or resistance exercise ≥ 2 times per week comparable to our intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy dose modifications | between baseline to 3rd/4th and 6th/8th treatment cycle or treatment switch. Cycle duration is 2 or 3 weeks.
  Number of patients requiring dose modifications (i.e. dose reductions, treatment delay, discontinuation or switch)
Progression free survival | between baseline and time to progression (up to 2 years)
  From date of randomization until the date of first documented progression

SECONDARY OUTCOMES:
NK-cell functionality | change from baseline to 6th treatment cycle or treatment switch (Cycle duration is 3 weeks)
  degranulation and cytotoxicity of NK-cells on peripheral blood mononuclear cells
Hospitalization | during treatment (6 treatment cycles of 3 weeks per cycle or 8 treatment cycles of 2 weeks per cycle)
  Number of patients requiring hospitalisation assessed from medical records
Treatment-related toxicity | change from baseline to 3rd/4th and 6th/8th treatment cycle or treatment switch (cycle duration is 2 or 3 weeks)
  severity of treatment-related toxicity assessed with the Common Terminology Criteria for Adverse Events
Aerobic fitness | change from baseline to 3rd/4th and 6th/8th treatment cycle or treatment switch (cycle duration is 2 or 3 weeks)
  Astrand-Rhyming test
Maximum short exercise capacity | change from baseline to 3rd/4th and 6th/8th treatment cycle or treatment switch (cycle duration is 2 or 3 weeks)
  Steep ramp test
Muscle strength | change from baseline to 3rd/4th and 6th/8th treatment cycle or treatment switch (cycle duration is 2 or 3 weeks)
  indirect 1 repetition maximum for leg press
Muscle mass | change from baseline to 3rd/4th and 6th/8th treatment cycle or treatment switch (cycle duration is 2 or 3 weeks)
  Computed Tomogrophy scans
Health-related quality of life | change from baseline to 3rd/4th and 6th/8th treatment cycle or treatment switch (cycle duration is 2 or 3 weeks)
  European Organization for Research and Treatment of Cancer Quality of Life Questionaire Core 30. Score from 0-100, higher scores indicate better functioning
Fatigue | change from baseline to 3rd/4th and 6th/8th treatment cycle or treatment switch (cycle duration is 2 or 3 weeks)
  European Organization for Research and Treatment of Cancer Quality of Life Questionaire- Fatigue 12. Score 0-100, higher scores indicate higher levels of fatigue
Resilience | change from baseline to 3rd/4th and 6th/8th treatment cycle or treatment switch (cycle duration is 2 or 3 weeks)
  Resilience Evaluation Scale, score 0-40, higher scores indicate better resilience
Empowerment | change from baseline to 3rd/4th and 6th/8th treatment cycle or treatment switch (cycle duration is 2 or 3 weeks)
  Self-efficacy-28, score 4-28, higher scores indicate better empowerment
Physical activity | change from baseline to 3rd/4th and 6th/8th treatment cycle or treatment switch (cycle duration is 2 or 3 weeks)
  Short QUestionnaire to ASsess Health enhancing physical activity, higher scores indicate higher physical activity levels

CONTACTS AND LOCATIONS:
Locations (13):
- Netherlands (13):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Flevoziekenhuis, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - Ziekenhuis Amstelland, Amstelveen
  - Amsterdam UMC, Amsterdam
  - Netherlands Cancer Institute, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Ziekenhuis Amphia, Breda
  - Catharina Ziekenhuis, Eindhoven
  - Spaarne Gasthuis, Hoofddorp
  - Radboudumc, Nijmegen
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - UMCU, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared via the POLARIS consortium see PROSPERO registry CRD42013003805 or paper: Buffart et al. Systematic Reviews 2013; 2: 75.

REFERENCES:
- [Derived] Brouwer CG, Tusscher MRT, de Roos BM, Gootjes EC, Buffart TE, Versteeg KS, Mast IH, Streppel MM, Werter IM, May AM, Verheul HMW, Buffart LM; AMICO Consortium. Experiences of patients with metastatic colorectal cancer participating in a supervised exercise intervention during chemotherapy. Support Care Cancer. 2025 Jan 8;33(2):82. doi: 10.1007/s00520-024-09101-1. PMID 39779537